CLINICAL TRIAL: NCT03602677
Title: Indocyanine Green Fluorescence Imaging in Prevention of Colorectal Anastomotic Leakage
Acronym: ICG-COLORAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oulu University Hospital (Other)
Collaborators: University of Oulu (Other); Central Finland Hospital District (Other); Tampere University Hospital (Other); Turku University Hospital (Other Government); Hospital District of Helsinki and Uusimaa (Other); Päijänne Tavastia Central Hospital (Other); Seinäjoki Central Hospital, Seinäjoki, Finland (Unknown)
Responsible Party: Principal Investigator, Olli Helminen, MD, PhD, Resident, Surgery, Oulu University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICG-COLORAL
Record Dates: First submitted 2018-03-25; First posted 2018-07-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Gastrointestinal Cancer; Gastrointestinal Neoplasms; Diverticulosis, Colonic; Gastrointestinal Disease
Keywords: Colorectal surgery; Anastomosis; Anastomosis leak; Fluorescence imaging
MeSH Terms: conditions — Colorectal Neoplasms; Gastrointestinal Neoplasms; Diverticulosis, Colonic; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG fluorescence imaging (Experimental): Colorectal surgery and anastomosis will be performed according to standard practice with the addition of intraoperative indocyanine green fluorescence imaging.
  Interventions: Device: ICG fluorescence imaging
- Standard procedure (No Intervention): Standard colorectal surgery and anastomosis.

INTERVENTIONS:
Device: ICG fluorescence imaging — The use of indocyanine green fluorescence imaging as an addition to standard surgical procedure.
  Arms: ICG fluorescence imaging

SUMMARY:
This is a randomized, controlled, parallel, multicenter trial to determine the difference in post-operative anastomotic leakages in colorectal surgery, where anastomosis perfusion is evaluated using indocyanine green fluorescence imaging as an addition to standard surgical practice compared to surgical practice alone.

ELIGIBILITY:
Inclusion Criteria:

* All consenting patients in the catchment area of participating hospitals who undergo elective colorectal surgery with planned primary anastomosis are eligible for this study.
* Of rectal cancer patients only those with pathology in the proximal third will be included in the study (defined by area proximal from peritoneal fold).

Exclusion Criteria:

* Emergent patients
* Patients with proven diverticular abscess and colonic fistulas are excluded
* Patients with planned open surgery are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1062 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Anastomosis leakage rate | 0 to 90 days

SECONDARY OUTCOMES:
Severity of anastomosis leakage | 0 to 90 days
  Grade A-C according to International Study Group of Rectal Cancer
Timing of anastomosis leakage | 0 to 90 days
  Days
Deep surgical site infections | 0 to 90 days
  Yes/no
Hospital readmission rate | 0 to 90 days
Reoperation rate | 0 to 90 days
30- and 90-day complications according to Clavien-Dindo Classification | 0 to 90 days
  Clavien-Dindo Score from Grade 0 (no complications) to Grade V (Death of a patient). Five grades and additionally Grade III and IV will be divided to a and b.
Operation time | 0-600 minutes
  Time from the start of the operation until the surgeon has ended the operation
Length of hospital stay | 0-365 days
  Day of the operation is considered the day 0
30- and 90-day mortality | 0 to 90 days
Time to first bowel movement | 0-30 days
  Postoperative day when the first bowel movement occurs
Time to first flatus | 0-30 days
  Postoperative day when the first flatus occurs
Hospital costs | 0 to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jyrki Kössi, MD, PhD, Principal Investigator — Päijänne Tavastia Central Hospital; Olli Helminen, MD, PhD, Principal Investigator — Oulu University Hospital, Oulu, Finland and Central Finland Central Hospital, Jyväskylä, Finland; Heikki Huhta, MD, PhD, Principal Investigator — Oulu University Hospital; Juha Rinne, MD, Principal Investigator — Päijänne Tavastia Central Hospital; Matti Kairaluoma, MD, PhD, Principal Investigator — Central Finland Central Hospital, Jyväskylä, Finland; Tero Rautio, MD, PhD, Principal Investigator — Oulu University Hospital
Locations (2):
- Finland (2):
  - Central Finland Central Hospital, Jyväskylä
  - Päijät Häme Central Hospital, Lahti

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinne JKA, Huhta H, Pinta T, Turunen A, Mattila A, Tahkola K, Helminen O, Ohtonen P, Rautio T, Kossi J. Indocyanine Green Fluorescence Imaging in Prevention of Colorectal Anastomotic Leakage: A Randomized Clinical Trial. JAMA Surg. 2025 May 1;160(5):486-493. doi: 10.1001/jamasurg.2025.0006. PMID 40042831

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT03602677/Prot_SAP_000.pdf